CLINICAL TRIAL: NCT07067749
Title: Treatment Expedition With MRI Processing and Optimization for Muscle Invasive Bladder Cancer
Acronym: TEMPO-MIBC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Simone Albisinni, Associate Professor of Urology, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 315.24CET2 ptv
Record Dates: First submitted 2025-06-10; First posted 2025-07-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Bladder Cancer Requiring Cystectomy; Bladder Carcinoma; Bladder Neoplasm; Muscle Invasive Bladder Cancer (MIBC)
Keywords: Muscle Invasive Bladder Cancer; VI-RADS; Bladder Magnetic Resonance Imaging; Cystectomy; TURBT; treatment expedition; cancer management optimisation; circulating tumour DNA
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging; Transurethral Resection of Bladder

STUDY DESIGN:
Intervention Model Description: Single centre, parallel, two-arm randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Management (Active Comparator): Patients enrolled in this arm will receive a flexible white light cistoscopy and concurrent cold-cup bladder tumour biopsy as part of the standard pathway at the sponsor Institution.
  They will be booked for TURBt and be managed according to international guidelines.
  If the pathology report of the TURBt will show muscle invasive bladder cancer, the clinical case will be discussed in the oncourological multidisciplinary board which will indicate the appropriate treatment.
  Treatment will be discussed with patients in a shared decision making context and booked.
  Management time monitoring will be conducted from the day of the cystoscopy until the day patients will receive the treatment indicated by the MDT.
  Interventions: Procedure: Transurethral resection of bladder tumour (TURBt); Genetic: Circulating tumour DNA levels assessment
- Simplified Management (Experimental): Patients enrolled in this arm will receive a flexible white light cistoscopy and concurrent cold-cup bladder tumour biopsy as part of the standard pathway at the sponsor Institution.
  They will be booked for bladder mpMRI through a dedicated service at the sponsor Institution to assess the suspiscion detrusor muscle invasion by the tumour.
  If the pathology report of the biopsy will show cancer and the mpMRI will confirm a high degree of suspicion for muscle invasive bladder cancer, the clinical case will be discussed in the oncourological multidisciplinary board which will indicate the appropriate treatment.
  Treatment will be discussed with patients in a shared decision making context and booked.
  Management time monitoring will be conducted from the day of the cystoscopy until the day patients will receive the treatment indicated by the MDT.
  Interventions: Diagnostic Test: multiparametric magnetic resonance imaging (mpMRI) of the bladder; Genetic: Circulating tumour DNA levels assessment

INTERVENTIONS:
Diagnostic Test: multiparametric magnetic resonance imaging (mpMRI) of the bladder — This study will investigate the role of bladder mpMRI as a tool to expedite treatment in patients with muscle invasive bladder cancer.
  mpMRIs will be investigated as a possible replacement of standard TURBt, a planned surgical procedure for cancer local staging.
  mpMRis will be reported according to the Vesical Imaging - Reporting and Data System Stanrdars (VI-RADS) to provide a score indicating probability of muscle invasion.
  Arms: Simplified Management
Procedure: Transurethral resection of bladder tumour (TURBt) — This is a planned endoscopic surgical procedure consisting in resection of the bladder tumour through a electrified loop manouvred with an endoscope. In muscle invasive bladder cancer, this procedure allows histological confirmation of presence of detrusor muscle invasion.
  Arms: Standard Management
Genetic: Circulating tumour DNA levels assessment — Blood samples will be collected from each enrolled patient at pre-planned time points:
  1. Cystoscopy, both arms
  2. mpMRI (experimental arm) or TURBt (control arm)
  3. Definite cancer treatment, both arms
  ctDNA levels will be measured on the collected blood samples.

SUMMARY:
The TEMPO-MIBC trial is a phase III, single-center, two-arm, randomized, controlled trial. Its primary objective is to evaluate the efficacy of a simplified diagnostic and treatment pathway for muscle-invasive bladder cancer (MIBC). This study investigates the role of multiparametric bladder MRI (mpMRI) in patients with biopsy proven cancer of the bladder with clinical features of detrusor muscle invasion. In the experimental arm, enrolled patients will receive a bladder mpMRI, if this exam will confirm the high suspicion of muscle invasion a conventional endoscopic transurethral resection of bladder tumour (TURBt) for staging purposes will be foregone and patients will immediately access the next step of their clinical management. Experimental arm outcomes will be compared to a control arm in which all enrolled patients will be receiving TURBt as part of the standard management of bladder cancer. The aim of this study is demonstrating a significant reduction of the time needed to offer patients the definitive treatment for their disease, possibly ensuring better long-term oncological outcomes.

A blood sample will be collected from each patient enrolled in the study at pre-planned time points to measure the levels of circulating tumour (ctDNA), a primer will be built from bladder cancer biopsies performed at enrolment. ctDNA has been shown to be a proxy measure of tumour burden and residual molecular disease after treatment. The ctDNA levels in the experimental arm will be compared to those of the control arm to investigate wether foregoing endoscopic resection of the tumour and reducing time to definitive cancer treatment might be associated to lower ctDNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of muscle invasive bladder cancer at cystoscopy and pre-cystoscopy imaging

Exclusion Criteria:

* Anticipated survival < 3 months due to comorbidities
* Pregnant patients
* Breastfeeding patients
* Previous chemotherapy within 6 weeks
* Previous radiotherapy withing 6 weeks
* Previous TURBt within 6 weeks
* Severe renal impairment (eGFR < 40 mL/min/1.73 m2)
* non MRI-compatible metal implants
* Claustrophobia
* Denial of written consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-08-15 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Time to definitive treatment | From the day of enrollment at baseline until the day of the start of definitive treatment for muscle invasive bladder cancer. Expected timeframe between 45 and 180 days.
  Time in days needed to complete the diagnostic pathway, multidisciplinary board discussion and finally offer the appropriate definitive treatment for muscle invasive bladder cancer: surgery, drugs, radiation, palliative care

SECONDARY OUTCOMES:
Concentration of ctDNA levels | Three specific time points: 1) Enrolment at baseline 2) During intervention (mpMRI or TURBt) 3) On the day of definitive treatment for muscle invasive cancer Expected timeframe 1 to 180 days
  ctDNA leves from blood samples collected at pre-planned time points in both arms
Cancer Specific Survival | through study completion, an average of 2 years
  Length of time from enrolment to the date of death from the disease.
Overall Survival | through study completion, an average of 2 years
  Length of time from enrolment to the date of death from any cause
Time to cancer recurrence | "through study completion, an average of 2 years".
  Length of time from enrolment to the date of clinically proven cancer recurrence
Number of procedure Related Complications | For 30 days following the procedure
  Monitoring of procedure related complications for TURBt and mpMRI

CONTACTS AND LOCATIONS:
Overall Officials: Simone Albisinni, MD, Phd, FEBU, Principal Investigator — Fondazione PTV Policlinico Tor Vergata
Locations (1):
- Policlinico Tor Vergata, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data to be released to other parties upon reasonable request to the Principal Investigatorand Local Ethics Board approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information available from study completion on August 2030 for 10 years
Access Criteria: Individual patient data to be released to other parties upon reasonable request to the Principal Investigator and Local Ethics Board approval